CLINICAL TRIAL: NCT00698646
Title: A 16 Week Multi-center, Randomized, Double-blind Study to Evaluate Efficacy and Safety of Valsartan/Hydrochlorothiazide (HCTZ) Combination Therapy Compared to Patients Initiated With Valsartan Monotherapy or Hydrochlorothiazide (HCTZ) Monotherapy in Very Elderly Patients With Essential Hypertension
Brief Title: Efficacy and Safety of Valsartan/Hydrochlorothiazide Combination Compared to Valsartan Monotherapy or Hydrochlorothiazide Monotherapy in Elderly (>70) With Mild-moderate Hypertension.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVAH631BUS08
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Results first posted 2010-12-15 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Hypertension
Keywords: Systolic blood pressure; Diastolic blood pressure; Valsartan; Hydrochlorothiazide
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Valsartan (Active Comparator): (patients initiated on valsartan)
  Interventions: Drug: Valsartan
- HCTZ (Active Comparator): (patients initiated on HCTZ)
  Interventions: Drug: HCTZ
- Valsartan + HCTZ (Experimental): (patients initiated on Valsartan+HCTZ)
  Interventions: Drug: Valsartan + HCTZ

INTERVENTIONS:
Drug: Valsartan + HCTZ — At week 0 patients received V+HCTZ 160+12.5 mg capsules. Subjects not at BP goal <140/90 mmHg were uptitrated to V+HCTZ 320+12.5 mg at week 4 and if needed to V+HCTZ 320+25 mg at week 8 or 12.
  Arms: Valsartan + HCTZ
Drug: Valsartan — At week 0 patients received Valsartan(V) 160 mg capsule. Subjects not at BP goal <140/90 mmHg were uptitrated to V+HCTZ 160+12.5 mg at week 4 and if needed to V+HCTZ 320+12.5 mg at week 8, and V+HCTZ 320+25 mg at week 12.
  Arms: Valsartan
Drug: HCTZ — At week 0 patients received HCTZ 12.5 mg capsule. Subjects not at BP goal <140/90 mmHg were uptitrated to V+HCTZ 160+12.5 mg at week 4 and if needed to V+HCTZ 320+12.5 mg at week 8, and V+HCTZ 320+25 mg at week 12.
  Arms: HCTZ

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of initial treatment therapy with valsartan/hydrochlorothiazide (HCTZ) versus the initial treatment therapy with monotherapies (valsartan or HCTZ) in the very elderly patients (greater than or equal to 70 years) with stage 1 or 2 hypertension

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years or older.
* Patients with hypertension prior to being randomized into study.
* Patients must have an office cuff MSSBP ≥ 140 and ≤ 200 mmHg systolic.
* Have the ability to communicate and comply with all study requirements.
* Provide written informed consent to participate in the study prior to any screening or study procedures.

Exclusion Criteria:

* Use of other investigational drugs within 30 days of enrollment.
* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
* Office blood pressure measured by office machine cuff with a mean of (3) MSDBP ≥ 120 mmHg at anytime during the screening / washout period.
* Patients taking 3 or more antihypertensive drugs and MSSBP ≥ 160 mmHg at the time of Visit 1.
* Other protocol-defined exclusion criteria may apply

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 384 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Investigative site, Birmingham, Alabama
  - Investigative site, Phoenix, Arizona
  - Investigative Site, Escondido, California
  - Investigative site, Fresno, California
  - Investigative site, Huntington Park, California
  - Investigative Sites, Pismo Beach, California
  - Investigative site, Miami, Florida
  - Investigative site, Ormond Beach, Florida
  - Investigative site, Conyers, Georgia
  - Investigative Site, Lexington, Kentucky
  - Investigative site, Portland, Maine
  - Investigative site, Las Vegas, Nevada
  - Investigative site, Buffalo, New York
  - Investigative site, Shelby, North Carolina
  - Investigative site, Carlisle, Ohio
  - Investigative site, Oklahoma City, Oklahoma
  - Investigative site, Erie, Pennsylvania
  - Investigative Site, Greer, South Carolina
  - Investigative Site, Taylors, South Carolina
  - Investigative site, St. George, Utah

REFERENCES:
- [Derived] Cushman WC, Duprez DA, Weintraub HS, Purkayastha D, Zappe D, Samuel R, Izzo JL Jr. Home and clinic blood pressure responses in elderly individuals with systolic hypertension. J Am Soc Hypertens. 2012 May-Jun;6(3):210-8. doi: 10.1016/j.jash.2012.03.001. PMID 22520932
- [Derived] Weintraub HS, Duprez DA, Cushman WC, Zappe DH, Purkayastha D, Samuel R, Izzo JL Jr. Antihypertensive response to thiazide diuretic or angiotensin receptor blocker in elderly hypertensives is not influenced by pretreatment plasma renin activity. Cardiovasc Drugs Ther. 2012 Apr;26(2):145-55. doi: 10.1007/s10557-011-6365-x. PMID 22311004
- [Derived] Izzo JL Jr, Weintraub HS, Duprez DA, Purkayastha D, Zappe D, Samuel R, Cushman WC. Treating systolic hypertension in the very elderly with valsartan-hydrochlorothiazide vs. either monotherapy: ValVET primary results. J Clin Hypertens (Greenwich). 2011 Oct;13(10):722-30. doi: 10.1111/j.1751-7176.2011.00498.x. Epub 2011 Jul 14. PMID 21974759
- [Derived] Duprez DA, Weintraub HS, Cushman WC, Purkayastha D, Zappe D, Samuel R, Izzo JL Jr. Effect of valsartan, hydrochlorothiazide, and their combination on 24-h ambulatory blood pressure response in elderly patients with systolic hypertension: a ValVET substudy. Blood Press Monit. 2011 Aug;16(4):186-96. doi: 10.1097/MBP.0b013e32834944e9. PMID 21747241
- See also: Click here for more information on the clinical study — http://www.novartisclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Valsartan: At week 0 patients received Valsartan 160 mg capsule. Subjects not at BP goal <140/90 mmHg were uptitrated to V+HCTZ 160+12.5 mg at week 4 and if needed to V+HCTZ 320+12.5 mg at week 8, and V+HCTZ 320+25 mg at week 12
Period: Overall Study
Arm/Group | Valsartan | HCTZ | Valsartan + HCTZ
Started | 128 | 128 | 128
Completed | 92 | 97 | 99
Not Completed | 36 | 31 | 29
Not completed — Adverse Event | 8 | 7 | 8
Not completed — Unsatisfactory Therapeutic Effect | 11 | 11 | 7
Not completed — Protocol Deviation | 6 | 2 | 3
Not completed — Withdrawal by Subject | 10 | 11 | 8
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Administrative problems | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan | HCTZ | Valsartan + HCTZ | Total
Number analyzed (Participants) | 128 | 128 | 128 | 384
Age Continuous [Mean (Standard Deviation); unit: years] | 77.7 (4.22) | 77.7 (4.80) | 77.2 (3.99) | 77.5 (4.34)
Age, Customized [Number; unit: participants]
  70-75 years | 41 | 41 | 44 | 126
  76-80 years | 60 | 56 | 65 | 181
  >80 years | 27 | 31 | 19 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 62 | 71 | 214
  Male | 47 | 66 | 57 | 170

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in Office Cuff Mean Sitting Systolic Blood Pressure (MSSBP)
Time Frame: Baseline and Week 4
Population: Intent to treat (ITT), Last observation carried forward
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Valsartan | HCTZ | Valsartan + HCTZ
Number analyzed (Participants) | 128 | 126 | 126
mm Hg
  Baseline | 166.2 (11.07) | 164.5 (11.84) | 164.5 (11.86)
  Week 4 | 157.5 (19.71) | 150.9 (18.41) | 147.1 (18.35)
  Change in MSSBP from Baseline to Week 4 | -8.6 (19.47) | -13.6 (16.81) | -17.3 (17.61)

2. Secondary Outcome: Change From Baseline to Week 4, 8, 12 and 16 in Office Cuff Mean Sitting Diastolic Blood Pressure (MSDBP)
Time Frame: Baseline and Weeks 4, 8, 12 and 16
Population: Intent to treat (ITT), Last observation carried forward
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Valsartan | HCTZ | Valsartan + HCTZ
Number analyzed (Participants) | 128 | 126 | 126
mm Hg
  Baseline | 84.9 (9.78) | 85.5 (9.09) | 84.8 (9.36)
  Week 4 | 81.0 (10.61) | 81.6 (10.97) | 77.8 (9.66)
  Change in MSDBP from Baseline to Week 4 | -3.9 (9.08) | -3.9 (10.24) | -7.1 (8.80)
  Week 8 | 78.3 (10.33) | 79.1 (11.97) | 76.5 (9.45)
  Change in MSDBP from Baseline to Week 8 | -6.6 (10.26) | -6.4 (10.72) | -8.4 (9.68)
  Week 12 | 77.6 (11.0) | 78.1 (11.42) | 75.4 (8.87)
  Change in MSDBP from Baseline to Week 12 | -7.3 (10.55) | -7.3 (10.75) | -9.5 (9.66)
  Week 16 | 77.8 (10.34) | 77.9 (11.66) | 76.6 (8.42)
  Change in MSDBP from Baseline to Week 16 | -7.1 (10.78) | -7.5 (10.76) | -8.3 (8.62)

3. Secondary Outcome: Change From Baseline to Weeks 8, 12 and 16 in Office Cuff Mean Sitting Systolic Blood Pressure (MSSBP)
Time Frame: Baseline and Weeks 8, 12, and 16
Population: Intent to treat (ITT), Last observation carried forward
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Valsartan | HCTZ | Valsartan + HCTZ
Number analyzed (Participants) | 128 | 126 | 126
mm Hg
  Baseline | 166.2 (11.07) | 164.5 (11.84) | 164.5 (11.86)
  Week 8 | 150.4 (20.29) | 147.4 (18.69) | 144.2 (19.93)
  Change in MSSBP from Baseline to Week 8 | -15.7 (20.43) | -17.1 (17.83) | -20.2 (19.12)
  Week 12 | 148.6 (21.45) | 145.1 (19.38) | 142.0 (18.78)
  Change in MSSBP from Baseline to Week 12 | -17.5 (21.16) | -19.4 (19.19) | -22.5 (19.52)
  Week 16 | 148.7 (20.06) | 144.9 (19.59) | 143.5 (18.69)
  Change in MSSBP from Baseline to Week 16 | -17.5 (19.62) | -19.7 (19.69) | -20.9 (18.49)

4. Secondary Outcome: Cumulative Percentage of Patients Achieving the Blood Pressure Control of < 140/90 mmHg
Description: Cumulative refers to achieving of blood pressure control before or at the corresponding visit.
Time Frame: Weeks 4, 8, 12 and 16
Population: Intent to treat (ITT)
Measure: Number; unit: Percentage of Participants
Arm/Group | Valsartan | HCTZ | Valsartan + HCTZ
Number analyzed (Participants) | 128 | 126 | 126
Percentage of Participants
  Week 4 | 25 | 37.3 | 49.21
  Week 8 | 40.63 | 50.79 | 63.49
  Week 12 | 50 | 61.11 | 69.05
  Week 16 | 55.47 | 66.67 | 72.22

5. Secondary Outcome: Cumulative Percentage of Patients Achieving Blood Pressure Goal (MSSBP < 140 mmHg)
Description: Cumulative refers to achieving blood pressure goal before or at the corresponding visit.
Time Frame: Weeks 4, 8, 12 and 16
Population: Intent to treat (ITT)
Measure: Number; unit: Percentage of Participants
Arm/Group | Valsartan | HCTZ | Valsartan + HCTZ
Number analyzed (Participants) | 128 | 126 | 126
Percentage of Participants
  Week 4 | 25 | 38.89 | 49.21
  Week 8 | 40.63 | 52.38 | 63.49
  Week 12 | 50 | 62.70 | 69.05
  Week 16 | 56.25 | 68.25 | 72.22

6. Secondary Outcome: Time in Weeks to Achieving the First Treatment Success (Defined as the Time of the First Achievement of the Target Blood Pressure Goal [MSSBP/MSDBP <140/90 mmHg])
Time Frame: During 16 weeks
Population: Intent to treat (ITT)
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Valsartan | HCTZ | Valsartan + HCTZ
Number analyzed (Participants) | 128 | 126 | 126
Weeks | 12.0 [8.0 to 12.0] | 8.0 [7.0 to 12.0] | 4.0 [3.0 to 8.0]

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Valsartan + HCTZ | HCTZ | Valsartan
Serious Adverse Events (participants affected / at risk) | 3/128 | 4/128 | 3/128
Other Adverse Events (participants affected / at risk) | 16/128 | 27/128 | 23/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan + HCTZ (N=128) | HCTZ (N=128) | Valsartan (N=128)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan + HCTZ (N=128) | HCTZ (N=128) | Valsartan (N=128)
Fatigue (General disorders) | 5 | 10 | 5
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 8
Dizziness (Nervous system disorders) | 5 | 8 | 9
Headache (Nervous system disorders) | 6 | 9 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.